CLINICAL TRIAL: NCT06791122
Title: A Multicenter, Pragmatic Study to Evaluate Clinical Effectiveness, Engagement With the Study App, Healthcare Resource Utilization, and Safety of an Investigational Digital Therapeutic (CT-155) in Patients With Experiential Negative Symptoms of Schizophrenia
Brief Title: A Prospective Cohort Study to Assess Clinical Effectiveness of an Investigational Digital Therapeutic (CT-155) in Patients With Experiential Negative Symptoms of Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1471-0002
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CT-155 treatment arm (Experimental)
  Interventions: Device: Digital therapeutic (CT-155)

INTERVENTIONS:
Device: Digital therapeutic (CT-155) — Digital therapeutic (CT-155) - in the form of a smartphone app

SUMMARY:
This study is open to people aged 18 years or older with schizophrenia. People can join the study if they are willing to use a smartphone app called CT-155. This app is being developed to help people with schizophrenia manage their negative symptoms.

The purpose of this study is to gather new information on CT-155. Researchers want to see how well it works, how well participants use the study app, and how it affects the use of health care services.

Participants use the app for 16 weeks. They may continue using it for another 16 weeks. During the study, participants continue with their normal treatment for schizophrenia. Participants are in the study for about a year. During this time, they visit the study site every 2 months.

During this study, doctors regularly check participants' schizophrenia symptoms and overall quality of life. Researchers may also compare the healthcare data of study participants with a similar group of people with schizophrenia who are not part of the study. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria

1. Has a primary diagnosis of schizophrenia using the diagnostic criteria for schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5 TR), and/or International Classification of Disease-10 (ICD-10) diagnosis code consistent with a schizophrenia diagnosis.
2. Has a Clinical Global Impression - Schizophrenia (CGI-SCH) negative symptoms score (item #2) ≥ 4 (moderately ill) at Screening.
3. 18 years of age or older at the time of informed consent.
4. Is willing and able to use CT-155 in English language regularly, to provide written informed consent to participate in the study and to be compliant with study-related assessments and activities.
5. Has outpatient treatment status at the time of screening, with no inpatient treatment for schizophrenia within 12 weeks prior to Screening.
6. Is on an antipsychotic medication(s) for at least 12 weeks prior to study entry.
7. Is the sole user of an iPhone with an iPhone operating system (iOS) 16+ or a smartphone with an Android operating system (OS) 12+ with a United States telephone number, and is willing to download and use the specified digital mobile application required by the protocol.
8. Is willing and able to receive SMS text messages and push notifications on their smartphone.

Further inclusion criteria apply.

Exclusion Criteria

1. Has a score of ≥3 (mildly ill) for CGI-SCH positive symptoms (item #1) at Screening.
2. Has active substance use disorder of any severity in the last 3 months, other than caffeine and nicotine. Patients are excluded if they fulfill criteria for moderate or severe substance use disorder for cannabis. Only mild substance use disorder for cannabis is allowed if considered by investigator to not impact ability of the patient to participate in the study.
3. Has suicidal ideation or behavior, as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS):

   * Patients with a "yes" response to either Items #4 or #5 on the C-SSRS Suicidal Ideation Item within the last 3 months (12 weeks) prior to screening, or at Screening.
   * Patients with a "yes" response on the C-SSRS Suicidal Behavior Items within the last 6 months (26 weeks) prior to screening or at Screening.
4. Patients who, in the opinion of the investigator, present a risk of suicide.
5. Is currently enrolled or has participated in the last 3 months (12 weeks) in a mental health related clinical study (interventional or observational).
6. Has participated in previous studies of CT-155 or CT-156.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
To assess the change from Baseline to Week 16 in negative symptoms severity, as assessed by the CGI-SCH negative symptoms item 2 among patients with schizophrenia using the investigational CT-155 Digital Therapeutic (DTx) | up to 16 weeks
  The Clinical Global Impression - Schizophrenia (CGI-SCH) contains 2 categories: severity of illness and degree of change.
  The severity of illness category evaluates the situation during the week prior to the assessment, while the degree of change category evaluates the change from the previous evaluation.
  Each category contains 5 different ratings (positive, negative, depressive, cognitive and global) that are evaluated using a seven-point ordinal scale (1 [Normal, not ill] - 7 [Among the most severely ill]) with higher ratings indicating more severe illness (severity of illness) or worsening of symptoms (degree of change).
To assess the change from Baseline to Week 16 in experiential negative symptoms (ENS), as assessed by the Motivation and Pleasure Scale Self-Report (MAP-SR) among patients with schizophrenia using the investigational CT-155 DTx | up to 16 weeks
  The MAP-SR is an 15-item self-report version of the Clinical Assessment Interview for Negative Symptoms Motivation and Pleasure subscale.
  Six items evaluate consummatory and anticipatory pleasure related to social and recreational or work domains; 3 items evaluate feelings and motivations to be around family, romantic partners, and friends; 6 items evaluate motivation and effort to engage in activities.
  All items are rated on a 5-point Likert scale (0 [not at all] - 4 [extreme pleasure]) with lower scores representing greater pathology.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Sun Valley Behavioral Med Center, Imperial, California
  - University of California San Diego, La Jolla, California
  - North Country Clinical Research Inc, Oceanside, California
  - ATP Clinical Research, Inc., Orange, California
  - NRC Research Institute, Orange, California
  - Stanford University Medical Center, Stanford, California
  - Collaborative Neuroscience Research, Torrance, California
  - CT Clinical Research, Cromwell, Connecticut
  - Galiz Research, Hialeah, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - University of Miami, Miami, Florida
  - Global Life Research Network, Miami, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Sheppard Pratt Physicians's Practice Association, Inc., Baltimore, Maryland
  - Center for Behavioral Health, LLC, Gaithersburg, Maryland
  - Boston Neurobehavioral Associates, Brookline, Massachusetts
  - University of Massachusetts - Worcester, Worcester, Massachusetts
  - Western Michigan University, Kalamazoo, Michigan
  - St. Charles Psychiatric Associates & Midwest Research Group, Saint Charles, Missouri
  - IMA Clinical Research Las Vegas, Las Vegas, Nevada
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Atrium Health, Charlotte, North Carolina
  - Rivus Wellness and Research Institute, Oklahoma City, Oklahoma
  - Psychiatric Consultants,PC, Franklin, Tennessee
  - Beaumont Psychiatry Clinic, Beaumont, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Salem VA Medical Center, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com